CLINICAL TRIAL: NCT04669860
Title: Evaluating the Bacterial and Fungal Microbiome in Patients With Calcium Oxalate Urolithiasis and Renal Cell Carcinoma.
Status: Suspended | Type: Observational
Why Stopped: lack of funding
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hemendra Shah, Professor of clinical Urology, University of Miami
Other Study IDs: 20200100
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Calcium Oxalate Urolithiasis; Renal Cell Carcinoma
Keywords: calcium oxalate stones; renal cell carcinoma; microbiome; urinary microbiome
MeSH Terms: conditions — Nephrolithiasis, Calcium Oxalate; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the microbiome of voided urine, bladder urine, stone fragments, and tissue from renal papillary biopsies in patients with CO stones.
  The microbiome of urine from the bladder, tissue from the renal tumor, and tissue from surrounding healthy renal tissue in patients with RCC
  Voided urine sample from healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- calcium oxalate urolithiasis group: Participants with CO urolithiasis scheduled for definitive endoscopic stone removal will be evaluated to identify bacterial and fungal microbiome in mid-stream voided urine sample, urine sample collected from the bladder, kidney stone fragment, and a renal papillae biopsy specimen.
- renal cell carcinoma group: Participants with RCC scheduled for definitive kidney removal surgery will be evaluated to identify bacterial and fungal microbiome in a catheterized urine specimen from the bladder, a biopsy of the tumor, and a biopsy of normal-appearing renal papillae specimen.
- healthy control group: The participants will provide a clean-catch voided midstream urine sample to identify bacterial and fungal microbiome.

SUMMARY:
The purpose of the study is to identify bacterial and fungal microbiome associated with calcium oxalate (CO) urolithiasis and renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

* Adults that are able to consent (≥ 18 years of age)
* No history of asymptomatic bacteriuria or Urinary Tract Infection within the past 1 month
* No history of coagulopathy and not on anticoagulant or antiplatelet medication at the time of surgery.
* For patients with urolithiasis, must not have a history of RCC
* For patients with RCC, must not have a history of urolithiasis
* Controls must have no history of stones, RCC, or urinary tract infection (within 1 month).
* For all participants, no antimicrobial treatment within the past month

Exclusion Criteria:

* Adults unable to consent
* For patients with urolithiasis, technical difficulty in taking renal papillae biopsy.
* History of urinary tract infection within the past 1 month
* History of coagulopathy and on anticoagulants or antiplatelets that could not be stopped perioperatively.
* Patients with nephrolithiasis and renal tumors with positive preoperative urine cultures- suggesting asymptomatic bacteriuria.
* For patients with urolithiasis, a history of RCC
* For patients with RCC, a history of urolithiasis
* Controls who have a history of stones, RCC, or urinary tract infection.
* For all participants, antimicrobial treatment within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy participants
  2. Participants with CO urolithiasis scheduled for endoscopic kidney stone removal surgery.
  3. Participants with RCC who are scheduled for kidney removal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Microbial community structure in patients with CO urolithiasis | Day 1
  Alpha and beta diversity, principal coordinate analysis, and phylogenetic trees of the bacterial and fungal microbial community from mid-stream voided urine sample, urine sample collected from the bladder, kidney stone fragment, and a renal papillae biopsy specimen.
Microbial community structure in patients with RCC | Day 1
  Alpha and beta diversity, principal coordinate analysis, and phylogenetic trees of the bacterial and fungal microbial community from catheterized urine specimen from the bladder, a biopsy of the tumor, and a biopsy of normal-appearing renal papillae specimen.
Microbial community structure in healthy participants | Day 1
  Alpha and beta diversity, principal coordinate analysis, and phylogenetic trees of the bacterial and fungal microbial community from clean-catch urine specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Hemendra N Shah, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No